CLINICAL TRIAL: NCT04833621
Title: Is Neuromuscular Electrical Stimulator Treatment in Sepsis/ Septic Shock Patients Protective in the Development of Intensive Care Unit Acquired Muscle Weakness (ICU-AW)?
Brief Title: Is NMES Treatment in Sepsis/ Septic Shock Patients Protective in Development of ICU-AW?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, GUNES COMBA CEBECI, RESIDENT, Ondokuz Mayıs University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01.02.2018 V:01
Record Dates: First submitted 2021-02-19; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Intensive Care Unit Acquired Weakness; Sepsis, Severe
Keywords: ICU-AW; NMES; sarcopenia; sepsis.
MeSH Terms: conditions — Sepsis; Sarcopenia

STUDY DESIGN:
Intervention Model Description: SINGLE CENTER, PROSPECTIVE, DOUBLE BLINDED
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES GROUP (Active Comparator): NMES TREATMENT AND PHYSICAL TREATMENT
  Interventions: Device: NMES GROUP
- CONTROL GROUP (Active Comparator): JUST PHYSICAL TREATMENT
  Interventions: Device: NMES GROUP

INTERVENTIONS:
Device: NMES GROUP — The effects of NMES and muscle strengthening and standard physiotherapy exercises on the development of ICU-AW were observed

SUMMARY:
Background: Sarcopenia (muscle weakness) characterized by a decrease in muscle mass, strength and performance is a condition that increases with old age. Sarcopenia can be seen in 5-13% of patients hospitalized in ICU where various treatment methods are used to prevent this weakness, the rate increases in patients with sepsis/ septic shock. Muscle treatment methods are used to prevent sarcopenia in similar patients hospitalized in ICU. It is predicted that "neuromuscular electrical stimulator-NMES" treatment may increase muscle mass and strength in patients who's can not be exercised actively. In this study, the contribution of NMES treatment to prevent the development of muscle weakness in patients with a diagnosis of sepsis/ septic shock followed in intensive care units (ICU) was evaluated.

DETAILED DESCRIPTION:
Background: Sarcopenia (muscle weakness) characterized by a decrease in muscle mass, strength and performance is a condition that increases with old age. Sarcopenia can be seen in 5-13% of patients hospitalized in ICU where various treatment methods are used to prevent this weakness, the rate increases in patients with sepsis/ septic shock. Muscle treatment methods are used to prevent sarcopenia in similar patients hospitalized in ICU. It is predicted that "neuromuscular electrical stimulator-NMES" treatment may increase muscle mass and strength in patients who's can not be exercised actively. In this study, the contribution of NMES treatment to prevent the development of muscle weakness in patients with a diagnosis of sepsis/ septic shock followed in intensive care units (ICU) was evaluated.

Patients and methods: In our single-center, prospective clinical study, 80 patients with a diagnosis of sepsis/ septic shock who were hospitalized in ICU were included. The effects of NMES and muscle strengthening and standard physiotherapy exercises on the development of ICU-AW were observed. The day when our patients were diagnosed with sepsis was recorded as the first day of the study. Anthropometric and ultrasonographic measurements of bilateral biceps brachii and bilateral rectus femoris muscles were recorded on the following days i.e. 3, 7, 14, 21, and 28. Sarcopenia was defined by anthropometric and ultrasonographic measurement, and all patient outcome data were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being in the Intensive Care Unit
* Over the age of 18
* Diagnosed with sepsis/ septic shock

Exclusion Criteria:

* Under the age of 18
* Pregnancy
* Having a cardiac pacemaker
* Amputated lower limbs
* Having severe venous insufficiency or major injuries to their lower extremities
* Having neuromuscular disease
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Effects of NMES treatment on ICU-AW development, anthropometric measurement, | 28 DAYS
  The measurements of the patients were recorded as anthropometric (arm circumference and thigh circumference) on the 1st, 3rd, 7th, 14th, 21st and 28th days. Arm circumference(centimeter) measurement was measured from the thickest part of the biceps muscle(centimeter) when the elbow was flexed and thigh circumference (centimeter) was measured anthropometrically with a tape measure (centimeter), 15 centimeter above the patella with the leg in extension.
Effects of NMES treatment on ICU-AW development, ultrasonographic measurement | on the 1st, 3rd, 7th, 14th, 21st and 28th days
  Using an ultrasound imaging device, the thickness of biceps brachii (cm^2) and rectus femoris muscles (cm^2) were measured ultrasonographically (at the same points of anthropometric measurements) with the linear probe.
Effects of NMES treatment on ICU-AW development, scoring systems. | on the 1st, 3rd, 7th, 14th, 21st and 28th days
  The muscle strength of the patients were evaluated according to the Medical Research Council (MRC) scoring.
Effects of NMES treatment on ICU-AW development, scoring systems. | on the 1st, 3rd, 7th, 14th, 21st and 28th days
  On the first day of the study, SOFA (Sequential Organ Failure Assessment) score,scoring systems were calculated for each patients.
Effects of NMES treatment on ICU-AW development, scoring systems. | first day
  On the first day of the study, qSOFA (quick Sequential Organ Failure Assessment) score scoring systems were calculated for each patients.
Effects of NMES treatment on ICU-AW development, scoring systems. | first day
  On the first day of the study, APACHE-II (Acute Physiology And Chronic Health Evaluation II) scoring systems were calculated for each patients.
Effects of NMES treatment on ICU-AW development, scoring systems. | 28 days
  When the follow-up was completed, duration of the ICU stay, intubated and/ or extubated days.
Effects of NMES treatment on ICU-AW development, scoring systems. | 28 days
  When the follow-up was completed, duration of the ICU stay, , last BMI (body mass index)(kg/m^2) were recorded.
Effects of NMES treatment on ICU-AW development, nutrition. | 28 days
  The diet of the patients were standardized by the dietitian.
height | first day and last day ( end of the 28th day)
  The height of the patients was calculated by measuring the knee height from many alternative height measurement methods. The measurement includes the length from the base of the foot to the anterior surface of the thigh while the lower extremity is flexed and is easily taken Chumlea et al. The equation created by the Chumlea method, known as the Chumlea method, is the most accurate equation used to estimate standing height from knee height. This method has been cross-validated for use in ICU patients. The original estimated equations are given.
  White Male Estimated height (cm) = (knee height (cm) × 1.88) + 71.85 White Female Estimated height (cm) = (knee height (cm) × 1.87) - (0.06 × age (y)) + 70.25
weight | first day and last day (end of the 28th day)
  We calculated the body weight of our patients by indirectly using the method of calculating body weight in bedridden patients.
  Age (Year) 6-18 Male : (Knee length (cm) x 0.68) + (Arm circumference (cm)x 2.64) -50.08 Female : (Knee (cm) x 0.77) + (Arm (cm) x 2.47) - 50.16
  19-59 Male : (Knee (cm) x 1.19) + (Arm (cm) x 3.21) -86.82 Female : (Knee (cm) x 1.01) + (Arm (cm) x 2.81) - 66.04
  60-80 Male : (Knee (cm) x 1.10) + (Arm (cm) x 3.07) -75.81 Female : (Knee (cm) x 1.09) + (Arm circumference(cm) x 2.68) - 65.51

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Faculty of Medicine, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided